CLINICAL TRIAL: NCT02640482
Title: A Randomized, Double-Blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus Genotype 2 Infection (ENDURANCE-2)
Brief Title: A Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Adults With Chronic Hepatitis C Virus (HCV) Genotype 2 Infection
Acronym: ENDURANCE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M15-464; 2015-002348-14 (EudraCT Number)
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Virus (HCV) Infection
Keywords: Treatment-Naive; Hepatitis C Virus Genotype 2; Sofosbuvir (SOF)-Experienced; Treatment-Experienced; Non-cirrhotic
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Infections | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A DB Active Drug (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks (double-blind [DB] treatment period)
  Interventions: Drug: ABT-493/ABT-530
- Arm B DB Placebo (Experimental): Placebo for ABT-493/ABT-530 QD for 12 weeks (DB treatment period)
  Interventions: Drug: Placebo for ABT-493/ABT-530
- Arm B OL Active Drug (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks (open-label [OL] treatment period)
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET
  Arms: Arm A DB Active Drug; Arm B OL Active Drug
Drug: Placebo for ABT-493/ABT-530 — tablet
  Arms: Arm B DB Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ABT-493/ABT-530 in adults with genotype 2 chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Screening laboratory result indicating hepatitis C virus (HCV) Genotype-2 (GT2) infection.
* Chronic HCV infection.
* Subject must be HCV treatment-naïve (subject had never received a single dose of any approved or investigational regimen) or had failed prior interferon (IFN) or pegylated-interferon (pegIFN) ± ribavirin (RBV) or sofosbuvir (SOF) + RBV ± pegIFN therapy.
* Subject must be non-cirrhotic.

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any excipient of the study drugs.
* Female who is pregnant, planning to become pregnant during the study, or breastfeeding; or male whose partner is pregnant or planning to become pregnant during the study.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
* HCV genotype performed during screening indicating coinfection with more than 1 HCV genotype.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Background] Asselah T, Kowdley KV, Zadeikis N, Wang S, Hassanein T, Horsmans Y, Colombo M, Calinas F, Aguilar H, de Ledinghen V, Mantry PS, Hezode C, Marinho RT, Agarwal K, Nevens F, Elkhashab M, Kort J, Liu R, Ng TI, Krishnan P, Lin CW, Mensa FJ. Efficacy of Glecaprevir/Pibrentasvir for 8 or 12 Weeks in Patients With Hepatitis C Virus Genotype 2, 4, 5, or 6 Infection Without Cirrhosis. Clin Gastroenterol Hepatol. 2018 Mar;16(3):417-426. doi: 10.1016/j.cgh.2017.09.027. Epub 2017 Sep 22. PMID 28951228
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety population: All participants who received at least one dose of study drug.
Pre-assignment Details: A total of 304 subjects were randomized and 302 subjects received at least 1 dose of study drug.
Groups:
- Arm B DB Placebo Then OL Active Drug: Placebo for ABT-493/ABT-530 QD for 12 weeks (DB treatment period) followed by ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks (open-label [OL] treatment period)
Period: Overall Study
Arm/Group | Arm A DB Active Drug | Arm B DB Placebo Then OL Active Drug
Started | 202 | 100
Completed | 199 | 100
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A DB Active Drug | Arm B DB Placebo Then OL Active Drug | Total
Number analyzed (Participants) | 202 | 100 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.77 (12.79) | 57.60 (12.04) | 57.04 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 55 | 159
  Male | 98 | 45 | 143

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Arm A DB Active Drug Excluding Prior SOF + Ribavirin (RBV) ± pegIFN Failures: Noninferiority Analysis
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of active study drug. The primary efficacy endpoint was the noninferiority of the percentage of participants who achieved SVR12 in Arm A Double Blind (DB) Active Drug excluding prior sofosbuvir (SOF) + ribavirin (RBV) ± pegylatedinterferon (pegIFN) failures compared with the historical control rate for patients treated with the current standard of care (SOF + RBV for 12 weeks).
Time Frame: 12 weeks after the last actual dose of active study drug
Population: All randomized participants who received at least one dose of study drug in Arm A DB excluding participants with prior SOF + RBV ± pegIFN failures.
Measure: Number; unit: percentage of participants
Groups:
- Arm A DB Active Drug: Arm A DB Active Drug: ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks (double-blind [DB] treatment period)
Arm/Group | Arm A DB Active Drug
Number analyzed (Participants) | 196
percentage of participants | 99.5
Statistical Analysis 1: Comparison: Arm A DB Active Drug; Based on a 2-sided significance level of 0.05 and an underlying rate of ≥96% in the Arm A (180 participants) provides >90% power to demonstrate noninferiority of ABT-493/ABT-530 to the historical rate for patients treated with the current standard of care (SOF + RBV for 12 weeks) (95%) (based on the normal approximation of using a single binomial proportion a one-sample test for superiority); Test type: Non-Inferiority — The noninferiority of the rate of sustained virologic response at 12 weeks after treatment for Arm A as compared with the historical rate for patients treated with the current standard of care (SOF + RBV for 12 weeks) was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 89% to achieve noninferiority; Percentage of Participants = 99.5, 95% CI 2-sided [98.5 to 100.0]

2. Secondary Outcome: Percentage of Participants With SVR12 in Arm A DB Active Drug Excluding Prior SOF + Ribavirin (RBV) ± pegIFN Failures: Superiority Analysis
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug. The secondary efficacy endpoint was the superiority of the percentage of participants who achieved SVR12 in Arm A Double Blind (DB) Active Drug excluding prior SOF + RBV ± pegIFN failures compared with the historical control rate for patients treated with the current standard of care (SOF + RBV for 12 weeks). As pre-specified in the study protocol, the primary outcome measure and the secondary outcome measure are not tested independently from each other. Rather, the two measures are ranked in a fixed sequential testing procedure that only if success was demonstrated for the primary outcome (i.e. non-inferiority test of Arm A SVR12 rate to the standard of care) did we test the first secondary outcome (i.e. superiority test of Arm A SVR12 rate to the standard of care).
Time Frame: 12 weeks after the last actual dose of active study drug
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm A DB Active Drug
Number analyzed (Participants) | 196
percentage of participants | 99.5
Statistical Analysis 1: Comparison: Arm A DB Active Drug; Based on a 2-sided significance level of 0.05 and an underlying rate of ≥96% in the Arm A (180 participants) provides >90% power to demonstrate superiority of ABT-493/ABT-530 to the historical rate for patients treated with the current standard of care (SOF + RBV for 12 weeks) (95%) (based on the normal approximation of a single binomial proportion using a one-sample test for superiority); Test type: Superiority — The superiority of the rate of sustained virologic response at 12 weeks after treatment for Arm A as compared with the historical rate for patients treated with the current standard of care (SOF + RBV for 12 weeks) was analyzed; the lower confidence bound of the 2-sided 95% confidence interval (95% CI) for the percentage of participants with sustained virologic response at 12 weeks after treatment must exceed 95% to achieve superiority; Percentage of Participants = 99.5, 95% CI 2-sided [98.5 to 100.0]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure in Arm A DB Active Drug Excluding Prior SOF + Ribavirin (RBV) ± pegIFN Failures
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value of post-baseline HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Up to Week 12 post baseline
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A DB Active Drug
Number analyzed (Participants) | 196
percentage of participants | 0.0 [0.0 to 1.9]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse in Arm A DB Active Drug Excluding Prior SOF + Ribavirin (RBV) ± pegIFN Failures
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of DB treatment and 12 weeks after the last dose of active study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: Between End of Treatment (Week 12) and 12 weeks after the last dose of Arm A DB active drug (up to Week 24)
Population: All randomized participants who received at least 1 dose of study drug in Arm A DB with HCV RNA < LLOQ at the final treatment visit who completed the DB treatment, excluding participants with prior SOF + RBV ± pegIFN failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A DB Active Drug
Number analyzed (Participants) | 195
percentage of participants | 0.0 [0.0 to 1.9]

5. Secondary Outcome: Percentage of Participants With SVR12 in Arm A DB Active Drug With Prior SOF + RBV ± pegIFN Failure
Description: SVR12 was defined as HCV RNA level <LLOQ 12 weeks after the last dose of active study drug.
Time Frame: 12 weeks after the last actual dose of active study drug
Population: All randomized participants who received at least one dose of study drug in Arm A DB with prior SOF + RBV ± pegIFN failures.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A DB Active Drug
Number analyzed (Participants) | 6
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks) for all participants in the double-blind (DB) period; TEAEs and TESAEs were also collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks) for all participants in the open-label (OL) period.
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug (or until prior to the first dose of open-label active drug for subjects who received DB placebo then OL active study drug) and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Arm A DB Active Drug | Arm B DB Placebo | Arm B OL Active Drug
Serious Adverse Events (participants affected / at risk) | 3/202 | 1/100 | 1/100
Other Adverse Events (participants affected / at risk) | 75/202 | 38/100 | 31/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A DB Active Drug (N=202) | Arm B DB Placebo (N=100) | Arm B OL Active Drug (N=100)
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A DB Active Drug (N=202) | Arm B DB Placebo (N=100) | Arm B OL Active Drug (N=100)
Diarrhoea (Gastrointestinal disorders) | 20 | 3 | 5
Nausea (Gastrointestinal disorders) | 15 | 4 | 8
Asthenia (General disorders) | 19 | 8 | 5
Fatigue (General disorders) | 23 | 10 | 5
Dizziness (Nervous system disorders) | 6 | 5 | 1
Headache (Nervous system disorders) | 24 | 12 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 6 | 5
Hypertension (Vascular disorders) | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.